CLINICAL TRIAL: NCT00666146
Title: Familial Schizophrenia and Spectrum Personality Disorders
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, MPRC, Gunvant Thaker, PI, University of Maryland, Baltimore
Other Study IDs: HP-00042566
Record Dates: First submitted 2008-04-21; First posted 2008-04-24 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Genetics; Eyetracking
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample for DNA extraction
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Case Families ( Family with a schizophrenia proband)
- 2: Control Families
- 3: Control subjects

SUMMARY:
We propose to recruit 150 case families (i.e., families with a schizophrenia proband), 150 control families, and 45 control subjects who exhibit schizophrenia spectrum personality symptoms in the absence of a family history of schizophrenia. Participants will undergo a number of clinical, electrophysiological, perceptual, and cognitive assessments. These data will be used to identify phenotypes likely to be associated with genetic risk for schizophrenia, and to determine how these phenotypes aggregate in families. Some of the analyses will focus on examining associations between candidate genes and these alternative phenotypes. Thus if we are not able to recruit relatives we may still collect these phenotypic data in probands and their genetic sample for future genotype/phenotype association studies. Testing procedures require a 10-12 hour time commitment and testing will be completed over 2 or more days. Participants will be asked to give a blood (or saliva if difficult to obtain blood sample for instance because of fear of blood draws), which will be stored for future genetic analyses.

DETAILED DESCRIPTION:
Specific aims of the proposed study are:

1. To test the hypothesis that abnormalities in predictive pursuit, antisaccade performance, working memory, visual attention (CPT), sensory gating (PPI and P50) and other measures of information processing mark the liability for schizophrenia. Secondly, we will examine the pattern of familial aggregation of these measures to determine whether observed deficits are likely to reflect genetic and/or environmental effects. The hypothesis will be supported if (a) the frequency of these neurophysiological deficits is higher in relatives of schizophrenic probands than in relatives of control probands; (b) the prevalence of neurophysiological abnormalities is higher in case relatives with SSP symptoms than in nonSSP case relatives; (c) risk is increased among case relatives of "affected" probands vs. case relatives of "unaffected" probands (i.e., risk in relatives of case probands who exhibit an abnormality vs. relatives of case probands who do not).
2. To test the hypothesis that some physiological deficits reflect a common underlying phenotype, while others mark independent aspects of disease risk. To test this hypothesis (a) we will examine correlation matrices (adjusted for within family correlation) for neurophysiological assessments among case relatives and control relatives. Factor structures in the two groups will be examined using exploratory factor analyses, followed by confirmatory factor analyses using validation samples of case/control relatives. Confirmatory Factor Analyses (CFA) will also be used to determine how factor solutions based on case/control relatives fit the data of case probands. (b) Factor scores for correlated measures will be derived and the familial risk for composite measures of neurophysiological functioning estimated using the methods described in Specific Aim 1. (c) Secondary within family analyses will be performed to estimate the heritability of derived factor scores and to determine whether patterns of familial correlations suggest a genetic or environmental cause.
3. To evaluate whether particular domains of psychopathology are marked by different putative phenotypic markers. We will specifically test the hypotheses that predictive pursuit, working memory, and sensory gating measures are more strongly associated with positive psychotic symptoms, while smooth pursuit initiation and processing speed measures are more strongly associated with primary negative symptoms. The relationships between clinical domains and other measures or clusters will be examined in an exploratory hypothesis-generating framework.
4. We propose to collect blood samples (or rarely saliva sample) from each participant to be stored for future association studies, as well as formal linkage analyses using phenotypes identified in specific aims 1 and 2.
5. We plan to examine how nicotine dependence may run in families and to examine if patterns of nicotine use may be related to a family history of schizophrenia. Participants will be asked about their smoking history and current smoking habits. Current smokers will be asked more specific questions about their smoking behaviors to estimate level of current nicotine dependence. It is hoped that this information will give us clues about why so many individuals with schizophrenia smoke.

ELIGIBILITY:
Inclusion Criteria:

* All male and female participants must be age 16 and above.
* Case probands will include individuals who meet DSM-IV criteria for schizophrenia or Research Diagnostic Criteria (RDC) for schizoaffective disorder.
* Control probands will include individuals matched with case probands with respect to age, gender, and county of residence who do not meet DSM-IV criteria for schizophrenia or other psychotic disorders.
* Case and control relatives will include all available and age-eligible first-degree relatives of identified case and control probands. Exception to this criterion will occur if we identify a schizophrenia proband family of large pedigree willing to participate, then we will include several generations of relatives (second, third or more degree) for subsequent linkage studies in a subgroup of our sample.
* SSP controls will include individuals recruited from the community who exhibit schizophrenia spectrum personality (SSP) traits in the absence of a personal or family history of psychotic illness.

Exclusion Criteria:

* Subjects under 16 years of age will be excluded.
* Subjects with serious medical, neuro-ophthalmological or neurological illness (e.g., cancer,seizure disorders,encephalopathy), current substance abuse or extensive history or drug dependence will be excluded, with the exception of subjects participating for clinical interview and blood sample only.
* Subjects with mental retardation will be excluded.
* Control probands and SSP controls who meet DSM-IV criteria for a psychotic illness, or have a family history of psychotic illness will be excluded.
* Schizophrenic patients who are judged to be incompetent to provide voluntary informed consent based on the ESC evaluation

Ages: 16 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: University of Maryland, Baltimore: Enrolling by Invitation
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2004-07; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Smooth pursuit eye movement measures; P50 gating; PPI; Cognitive measures; P300 component evoked potential; genetic markers | 12-16 hours

CONTACTS AND LOCATIONS:
Overall Officials: James Gold, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (3):
- United States (3):
  - Community Mental Health Centers, Baltimore, Maryland
  - VA Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Catonsville, Maryland

IPD SHARING:
Plan to Share IPD: No